CLINICAL TRIAL: NCT06856889
Title: Evaluation of the Value of Systematic Ultrasound in the Initial Assessment of Ankle Sprain on Functional Prognosis at 3 Months in the General Population: Pilot Observational Study (PFEEC)
Brief Title: Systematic Ultrasound in the Initial Assessment of Ankle Sprain
Acronym: PFEEC
Status: Recruiting | Type: Observational
Sponsor: Hopital Nord Franche-Comte (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-12-PFEEC
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Ankle Sprain
Keywords: ultrasound scan
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control group: no ultrasound scan
- Experimental groupe: ultrasound scan

SUMMARY:
Ankle sprains are the most frequently encountered trauma in emergency and general medicine. Lateral ankle sprain injuries have the highest relapse rate of all musculoskeletal injuries of the lower limbs. Optimal initial management is essential for a successful return to previous condition, with the aim of preventing chronic ankle instability, chronic pain, stiffness or recurrence. One of the 13 physicians at our facility routinely performs an ultrasound routinely scan during the second consultation to assess the severity of the sprain. We would therefore like to evaluate whether the performance of this examination at the time of clinical reassessment is associated with a better prognosis at 3 months post-trauma.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ankle sprain made during a preliminary prior consultation
* Patients undergoing re-evaluation of sprain severity, between D3 and D6 of trauma

Exclusion Criteria:

* Medial sprain
* Sprain recurrence <6 months
* Age < 15 years
* Radiographic fracture confirmed on an X-ray performed between initial diagnosis and re-evaluation visit
* History of hyperlaxity syndrome

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with ankle sprain
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2025-11-26 (Estimated); Study Completion 2025-11-26 (Estimated)

PRIMARY OUTCOMES:
Value of systematic ultrasound in the initial assessment of ankle sprains on patients' quality of life and sporting activities at 3 months post-injury trauma. | 3 months
  Comparison of ankle-specific quality of life in terms of activities of daily living and sporting activities. This criterion will be measured using the FAAM (Foot and Ankle Ability Measure), a specific questionnaire functional evaluation of the ankle in these activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Maison Médicale des Bords de Seille, Bletterans, France

IPD SHARING:
Plan to Share IPD: No